## Developing an Integrative, Recovery Based, Post-Acute COVID-19 Syndrome (PACS) Psychotherapeutic Intervention, "PACS Coping and Recovery"

**Funding Agency:** Rehabilitation Research and Development Service (RR&D) Small Projects in Rehabilitation Research (SPiRE).

NCT05453201

June 1, 2024

## **JJPVAMC**

PI: Marianne Goodman MD Co-I: Yosef Sokol PhD Co-I: Emily Edwards PhD

Co-I: Brittany Stevenson PhD

All statistical analyses were conducted using the RStudio (version 4.4.2). Item-level missingness (< 0.5% item-level observations) was handled with participant-mean imputation. Little's (1988) missing completely at random (MCAR) test was not significant (p > .05) indicating that the data were missing at random. Paired-sample t-tests were used to examine changes in primary and secondary outcomes from pre- to post-treatment. Paired Wilcoxon tests were used when the Shapiro-Wilk test was significant (p < .05). The significance level was set at p < .05 for all analyses.